CLINICAL TRIAL: NCT01445899
Title: An Open-Label Dose Escalation Study of PF-04523655 (Stratum I) Combined With a Prospective, Randomized, Double-Masked, Multi-Center, Controlled Study (Stratum II) Evaluating the Efficacy and Safety of PF-04523655 Alone and in Combination With Ranibizumab Versus Ranibizumab Alone in Diabetic Macular Edema (MATISSE STUDY)
Brief Title: PF-04523655 Dose Escalation Study, and Evaluation of PF-04523655 With/Without Ranibizumab in Diabetic Macular Edema (DME)
Acronym: MATISSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QRK202; 2011-004157-66 (EudraCT Number)
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Choroidal Neovascularization; Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Choroidal Neovascularization; Diabetic Retinopathy | interventions — PF-04523655; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PF-04523655 (Stratum II) (Experimental): Stratum II, 6 monthly injections of PF-04523655 only
  Interventions: Drug: PF-04523655 (Stratum II)
- PF-04523655 and ranibizumab (Experimental): Stratum II, 6 monthly injections of PF-0423655 and ranibizumab administered in combination
  Interventions: Drug: ranibizumab; Drug: PF-04523655 (Stratum II)
- ranibizumab (Active Comparator): Stratum II, 6 monthly IVT injections of ranibizumab only
  Interventions: Drug: ranibizumab
- PF-04523655 (Stratum I) (Experimental): Stratum I
  Interventions: Drug: PF-04523655 (Stratum I)

INTERVENTIONS:
Drug: PF-04523655 (Stratum I) — PF-04523655 (a small interfering RNA) - a single IVT injection
  Other Names: PF-655
  Arms: PF-04523655 (Stratum I)
Drug: ranibizumab — 6 monthly IVT injections of ranibizumab (Stratum II)
  Other Names: Lucentis
  Arms: PF-04523655 and ranibizumab; ranibizumab
Drug: PF-04523655 (Stratum II) — 6 monthly IVT injections of PF-04523655 (a small interfering RNA)
  Other Names: PF-655
  Arms: PF-04523655 (Stratum II); PF-04523655 and ranibizumab

SUMMARY:
This is a two-part study. The first part (Stratum I) is an open-label, dose escalation, safety, tolerability and pharmacokinetic study, where active study drug (PF-04523655) will be given to all patients who participate. Stratum I will determine the maximum tolerated dose and any dose-limiting toxicities. The second part (Stratum II) is a prospectively randomized, multi-center, double-masked, dose ranging study evaluating the efficacy and safety of PF-04523655 alone and in combination with ranibizumab versus ranibizumab alone in patients with DME.

DETAILED DESCRIPTION:
Patients will be enrolled concurrently according to one of two sets of criteria designated as Stratum I and Stratum II.

1. Stratum I will enroll up to 24 subjects with low vision, inclusive of possible intermediate doses, in up to 4 cohorts of 3-6 evaluable subjects.
2. Stratum II will enroll approximately 240 subjects with DME 1:1:1:1 in up to 4 cohorts of 60 evaluable subjects.

ELIGIBILITY:
Key Stratum I Inclusion Criteria:

1. Visual acuity in the study eye ≤ 20/200.
2. Low visual acuity is the result of an irreversible condition affecting the posterior segment of the study eye.

Key Stratum I Exclusion Criteria:

1. History of vitrectomy.
2. History of IVT injection in study eye within last 6 months.
3. History of vitreous hemorrhage, retinal detachment, or invasive trauma in study eye.
4. History of uveitis or endophthalmitis in either eye.
5. Any active inflammatory condition in study eye.
6. Received any drugs known to cause optic nerve or retinal toxicity within 14 days prior to dosing.
7. Any medical condition, concomitant therapy or previous incisional or laser surgery that, in the opinion of the Investigator, would preclude IVT injection in the study eye.
8. Intraocular pressure in either eye ≥25 mmHg on maximal medication.
9. Cataract surgery and laser corneal surgery within 3 months prior to dosing in the study eye and all other intraocular surgeries at any time.
10. Participation in a concurrent interventional study within 30 days prior to dosing.

Key Stratum II Inclusion Criteria:

1. History of diabetes mellitus (Type 1 or Type 2).
2. Retinal thickening secondary to the edema caused by diabetes mellitus.
3. Best corrected visual acuity (BCVA) of 20/40 or worse and up to 20/320 or better in the study eye at Screening.
4. Standard of care treatment for DME can be withheld for at least 90 days after the subject has enrolled in the study (study eye only).

Key Stratum II Exclusion Criteria:

1. History of panretinal photocoagulation within 6 months or macular laser photocoagulation within 3 months of prior to dosing in the study eye.
2. Any IVT injection therapy performed in the study eye within 3 months prior to dosing.
3. Iris neovascularization, vitreous hemorrhage, tractional retinal detachment, vitreomacular traction, clinically significant epiretinal membrane or clinically significant preretinal fibrosis involving the macula in the study eye.
4. History of vitreoretinal surgery or incisional glaucoma surgery in the study eye.
5. Prior intraocular surgery or corneal laser surgery, performed within 3 months prior to dosing in the study eye.
6. Received any drugs known to cause optic nerve or retinal toxicity within 14 days prior to dosing.
7. High risk (in the opinion of the Investigator) proliferative diabetic retinopathy (PDR) in the study eye.
8. Current infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
9. Monocular subjects.
10. History of idiopathic or autoimmune uveitis in either eye.
11. Aphakia or absence of the posterior capsule in the study eye.
12. Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema.
13. Uncontrolled glaucoma in either eye.
14. Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia.
15. Use of corticosteroids that, in the Investigator's opinion, may change the status of the subject's diabetic retinopathy in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and dose-limiting toxicities (Stratum I) | 6 months post-injection
  - To determine the safety and dose-limiting toxicities of a single intravitreal (IVT) injection of PF-04523655 in subjects with low vision
Pharmacokinetics (Stratum I) | 6 months post-injection
  - To determine the pharmacokinetics (PK) of a single IVT injection of PF-04523655 in subjects with low vision
Safety and tolerability (Stratum II) | 30 days after the last injection
  - To evaluate the safety and tolerability of PF-04523655 alone and in combination with ranibizumab in subjects with diabetic macular edema (DME)
Efficacy (Stratum II) | 30 days after the last injection
  - To evaluate the ability of PF-04523655 alone and in combination with ranibizumab to improve visual acuity compared to ranibizumab alone in subjects with DME

SECONDARY OUTCOMES:
Anatomical changes in retina and retinal nerve fiber layer morphology (Stratum II) | 30 days after the last injection
  - To evaluate the anatomical changes in retina and retinal nerve fiber layer (RNFL) morphology following administration of PF-04523655 alone and in combination with ranibizumab compared to ranibizumab alone by fundus photography (FP) and spectral domain optical coherence tomography (SD-OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, MD, Study Director — Quark Pharmaceuticals
Locations (51):
- United States (20):
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Retina Institute of California, Arcadia, California
  - Retina-Vitreous Associates, Beverly Hills, California
  - Retina Diagnostic Center, Campbell, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Orange County Reina Medical Group, Santa Ana, California
  - MedEye Associates, Miami, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Thomas A. Cuilla, MD, PC at Midwest Eye Institute, Indianapolis, Indiana
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - Retina Vitreous Center, Toms River, New Jersey
  - Southeast Clinical Research Associates, LLC, Charlotte, North Carolina
  - Black Hills Regioinal Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Center, Austin, Texas
  - Retinal Consultants of Houston, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retinal Institute of Virginia, Richmond, Virginia
- Belgium (2):
  - University Hospital Ghent, Ghent, Belgium
  - Brugmann Ziekenhuis, Laken, Belgium
- Czechia (4):
  - Fakultni nemocnice Brno, Brno, Czech Republic
  - Fakultní nemocnice Hradec Kralove, Kralove, Czech Republic
  - Fakultní nemocnice Ostrava, Ostrava, Czech Republic
  - GEMINI oční centrum, a.s, Zlín, Czech Republic
- Germany (5):
  - Augenärzte Gemeinschaftspraxis Ahaus-Gronau-Lingen-Münster-Bad Bentheim, Ahaus, Germany
  - Augenklinik Klinikum Darmstadt, Darmstadt, Germany
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen, Germany
  - Klinik und Poliklinik für Augenheilkunde Klinikum rechts der Isar, München, Germany
  - Augenklinik am St. Franziskus-Hospital Muenster, Münster, Germany
- Israel (9):
  - Soroka University Medical Center, Beersheba, Israel
  - Bnai Zion Medical Center, Haifa, Israel
  - Meir Medical Center, Kfar Saba, Israel
  - The Chaim Sheba Medical Center, Tel Litwinsky, Israel
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Ẕerifin
- Poland (4):
  - Oftalmika, Bydgoszcz, Poland
  - Szpital Specjalistyczny Nr 1 w Bytomiu, Bytom, Poland
  - Profesorskie Centrum Okulistyki, Hipermarket Tesco, Gdansk, Poland
  - Spectrum OOK, Wroclaw, Poland
- United Kingdom (7):
  - Southamptom Eye Unit, Southampton Hospital, Shirley, Southampton
  - Frimley Park Hospital NHS Foundation Trust, Frimley, Surrey
  - Eye and Ear Clinicl, The Royal Victoria Hospital, Belfast, United Kingdom
  - Bristol Eye Hospital, Bristol, United Kingdom
  - St. James University Hospital, Leeds, United Kingdom
  - Moorfields Eye Hospital, London, United Kingdom
  - Royal Hallamshire Hospital, Eye Department, Sheffield, United Kingdom